CLINICAL TRIAL: NCT03095469
Title: Effects of Dexmedetomidine on Patients With Coronary Heart Disease After Percutaneous Coronary Intervention:A Double-Blinded, Randomised Controlled Trial
Brief Title: Effects of Dexmedetomidine on Patients With Coronary Heart Disease After Percutaneous Coronary Intervention
Acronym: EODOPWCHD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJTU1AF-CRF-2016T-09
Record Dates: First submitted 2017-02-26; First posted 2017-03-29 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Heart Injuries
MeSH Terms: conditions — Heart Injuries | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: coronary artery disease patients with anxiety who receive selective PCI
Who Masked: Participant, Care Provider, Investigator
Masking Description: all of the participants, operators, investigators and outcomes assessors don't know the grouping situation before the study finished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): when the operation begin,dexmedetomidine will be pumped at 0.4μg/kg•h for 15 minutes ,then reduce the dose to 0.2μg/kg•h until 24 h after PCI.
  Interventions: Drug: Dexmedetomidine
- control group (Placebo Comparator): 0.9%NaCl solution 0.1ml/kg•h when the operation begin and stopped until 24 h after PCI.
  Interventions: Drug: 0.9%NaCl solution

INTERVENTIONS:
Drug: Dexmedetomidine — when the operation begin,dexmedetomidine will be pumped at 0.4μg/kg•h for 15 minutes ,then reduce the dose to 0.2μg/kg•h until 24h after PCI.
  Other Names: Dexmedetomidine Injection
  Arms: study group
Drug: 0.9%NaCl solution — when the operation begin,0.9%NaCl solution will be pumped at 0.1ml/kg•h until 24h after PCI.
  Other Names: Other Name: normal saline
  Arms: control group

SUMMARY:
Coronary heart disease has a high incidence and high death rate. Percutaneous coronary intervention (PCI) is an important method for the treatment of coronary heart disease (CHD). However, PCI may cause myocardial cell injury and myocardial infarction 4 Type(MI4a, Type 4 a myocardial infarction related to PCI). Dexmedetomidine(Dex) is the only anesthetic which has sedative and analgesic effects. Dex currently has been widely used in perioperative management of various surgical.This study intends to verify the effect of heart protection of Dex in perioperative.

DETAILED DESCRIPTION:
Participants will be randomly assigned, in a 1:1 ratio, to receive Dexmedetomidine or control (0.9 %Sodium Chloride Solution,0.9%NaCl). The randomization sequence will be computer-generated, and randomization will be performed in blocks and will be stratified according to participating center. Dexmedetomidine and 0.9 % NaCl solution will be transfused when the operation began, ending 24 hours after the surgery. Troponin I level(but are not limited to these data) at pre-operation and 3h, 6h,12h, 24h, 48h after PCI will be recorded. At the same time, other dates will be recorded.The participation of each patient is scheduled for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* the patients were coincided to CHD combined with depression and anxiety according to diagnostic standard of World Health Organization(WHO)who need receive selective PCI in the First Affiliated Hospital of Xi'an Jiaotong University;
* people aged over 18;
* patients who will undergo PCI with Hamilton Anxiety scale of 14 points or more.

Exclusion Criteria:

* severe comorbidity history;
* coronary stenosis less than 70%;
* severe cardiac dysfunction;
* central nervous system disease;
* troponin I levels have rised before entering the hospital;
* pregnant woman；
* history of mental disorders;
* alcoholic and long-term use of sedatives and opioids history;
* drug allergy history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08-20 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of myocardial infarction type 4a (MI4a) | detect serum TnI level before and 3h、6h、12h、24h、48h after PCI
  serum troponin(TnI) values at 48h after PCI is an important indicator for diagnosis of acute myocardial injury myocardial damage when troponin I lever rise.

SECONDARY OUTCOMES:
post-procedural cardiac function | once 3 months for 6 months after PCI
  Echocardiographic results can reflect cardiac function.Echocardiography index include left ventricular ejection fraction(LVEF),left ventricular end-diastolic diameter (LVEDD), left ventricular end-diastolic volume (LVEDV) and stroke volume (SV),doppler mitral flow E/A ratio(E/A).
major adverse cardiac events(MACEs) | once 3 months for 12 months after PCI
  MACEs' incidence reflects the incidence of MI4a
systemic inflammatory markers | before and 1 week after PCI
  systemic inflammatory markers can reflect the situation of cardiac injures,like tumor necrosis factor alpha(TNF-α),interleukin-6(IL-6),interleukin-8(IL-8),high-sensitivity C-reactive protein(hs-CRP).

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, PHD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- the 1st affiliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided